CLINICAL TRIAL: NCT02769676
Title: A Comparison of Short Interval vs. Routine Postpartum Visit on Contraceptive Initiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201512058
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3-week visit (Experimental): Participants randomized to this arm will receive an additional visit at 3-weeks postpartum
  Interventions: Other: 3-week visit
- usual care (Active Comparator): Participants randomized to this arm will receive usual postpartum care, including the standard timing for a postpartum visit.
  Interventions: Other: usual care

INTERVENTIONS:
Other: 3-week visit — The intervention will be an additional visit to the usual postpartum care provider at 3-weeks postpartum.
  Arms: 3-week visit
Other: usual care — Participants in the usual care arm will receive no additional interventions.
  Arms: usual care

SUMMARY:
The current postpartum care model of a single visit 4-6 weeks after delivery does not optimally address contraceptive needs. By this visit, many women have resumed sexual activity, potentially putting them at risk for unintended and rapid repeat pregnancy. In addition, many women with pregnancy-related Medicaid lose insurance coverage at this time, making it difficult to obtain long-acting reversible contraception (LARC) if desired. Therefore, an earlier postpartum visit may remove barriers to improve access to LARC thereby, reducing unintended and rapid repeat pregnancy. Our primary objective is to determine whether an additional 3-week postpartum visit, compared to usual postpartum care, will affect the initiation of LARC by 6 weeks postpartum.

DETAILED DESCRIPTION:
Our primary objective is to determine whether an additional 3-week postpartum visit, compared to usual postpartum care, will affect the initiation of LARC by 6 weeks postpartum. Our secondary outcomes include: 1) desired method of postpartum contraception; 2) continuation and satisfaction with contraception; and 3) incidence of rapid repeat and unintended pregnancy at 12 months. We will also measure attendance and satisfaction with 3- compared to 6-week postpartum visits.We will perform a two-arm randomized controlled trial (RCT). Women will be randomized to routine postpartum follow-up compared to two postpartum visits; one at 3 weeks and one at 6 weeks, with initiation of contraception at the 3-week visit as indicated. Women will be recruited from the postpartum service of Barnes-Jewish Hospital and all women will receive structured comprehensive counseling (adapted from the CHOICE Project Model) prior to discharge from the hospital. Postpartum visits will occur at our outpatient ambulatory clinic sites. Participants will complete in-person surveys at baseline and at each visit, and telephone surveys at 6- and 12-months postpartum. Planned recruitment will be 200 women based on a 2-fold increase in LARC initiation in the intervention group compared to control group (40% vs. 20% initiation rate).

ELIGIBILITY:
Inclusion Criteria:

* Delivered at Barnes-Jewish Hospital
* Receiving postpartum care at resident clinic

Exclusion Criteria:

* Received LARC, sterilization, or hysterectomy
* Abortion, stillbirth, or neonatal death
* Non-English speaking
* Unable to comply with follow-up

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2016-05; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Initiation of LARC by time of standard postpartum visit | 4-8 weeks postpartum
  Initiation of LARC method

SECONDARY OUTCOMES:
Contraceptive use at 6 & 12 months | 6 & 12 months postpartum
  Use of contraception
Unintended rapid-repeat pregnancy | 12 months postpartum
  Incidence of an unintended rapid-repeat pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Bernard, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yonemoto N, Nagai S, Mori R. Schedules for home visits in the early postpartum period. Cochrane Database Syst Rev. 2021 Jul 21;7(7):CD009326. doi: 10.1002/14651858.CD009326.pub4. PMID 34286512
- [Derived] Bernard C, Wan L, Peipert JF, Madden T. Comparison of an additional early visit to routine postpartum care on initiation of long-acting reversible contraception: A randomized trial. Contraception. 2018 Sep;98(3):223-227. doi: 10.1016/j.contraception.2018.05.010. Epub 2018 May 18. PMID 29778586